CLINICAL TRIAL: NCT06057610
Title: A Phase III Multicenter, Randomized, Open-label, Active-Controlled Study of SHR-A1811 With or Without Pertuzumab Versus Trastuzumab, Pertuzumab and Docetaxel in HER2-Positive Recurrent or Metastatic Breast Cancer
Brief Title: A Phase III Study of SHR-A1811 Injection With or Without Pertuzumab in HER2-Positive Recurrent or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-307
Record Dates: First submitted 2023-09-11; First posted 2023-09-28 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HER2-PositiveRecurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: SHR-A1811 Injection (Experimental)
  Interventions: Drug: SHR-A1811 Injection
- Treatment group B: SHR-A1811 Injection and Pertuzumab Injection (Experimental)
  Interventions: Drug: SHR-A1811 Injection ； Pertuzumab Injection
- Treatment group C: Trastuzumab Injection, Pertuzumab Injection and Docetaxel Injection (Active Comparator)
  Interventions: Drug: Trastuzumab Injection；Pertuzumab Injection ； Docetaxel Injection

INTERVENTIONS:
Drug: SHR-A1811 Injection — SHR-A1811 Injection
  Arms: Treatment group A: SHR-A1811 Injection
Drug: SHR-A1811 Injection ； Pertuzumab Injection — SHR-A1811 Injection ； Pertuzumab Injection
  Arms: Treatment group B: SHR-A1811 Injection and Pertuzumab Injection
Drug: Trastuzumab Injection；Pertuzumab Injection ； Docetaxel Injection — Trastuzumab Injection；Pertuzumab Injection ； Docetaxel Injection
  Arms: Treatment group C: Trastuzumab Injection, Pertuzumab Injection and Docetaxel Injection

SUMMARY:
To evaluate the efficacy and safety of SHR-A1811 with or without pertuzumab versus trastuzumab, pertuzumab and docetaxel in HER2-Positive Recurrent or Metastatic Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 (inclusive)
2. HER2 positive (IHC3+ or ISH+) unresectable or metastatic breast cancer confirmed by histology or cytology.
3. ECOG score is 0 or 1
4. An expected survival of ≥ 12 weeks
5. At least one measurable lesion according to RECIST v1.1 criteria
6. Have adequate renal and hepatic function
7. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. Have other malignancies within the past 5 years
2. Active central nervous system metastasis without surgery or radiotherapy
3. In (neoadjuvant) adjuvant therapy phase, the interval from the end of systemic therapy (excluding endocrine therapy) to the detection of recurrence/metastasis ≤12 months
4. Presence with uncontrollable third space effusion
5. Have undergone other anti-tumor treatment within 4 weeks before the first dose
6. A history of immune deficiency
7. Clinically significant cardiovascular disorders
8. Known or suspected interstitial lung disease
9. The toxicity from previous anti-tumor treatment has not recovered to ≤ grade I
10. Known hereditary or acquired bleeding tendency
11. Active hepatitis and liver cirrhosis
12. Presence of other serious physical or mental diseases or laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival by Blinded Independent Central Review | from first dose to disease progression, or death, whichever comes first, up to 3 years

SECONDARY OUTCOMES:
Progression Free Survival by investigators | from first dose to disease progression, or death, whichever comes first, up to 3 years
Overall Survival | from first dose to death, up to 6 years
Objective Response Rate | from first dose to disease progression or death, whichever comes first, up to 3 years
Duration of response | from first dose to disease progression or death, whichever comes first, up to 3 years
AE | from Day1 to 40 or 90 days after last dose
Incidence and severity of serious adverse events (SAE) | from Day1 to 40 or 90 days after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided